CLINICAL TRIAL: NCT01845233
Title: Monitoring of Non-invasive Ventilation
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); Trondheim University Hospital (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1142(REK)
Record Dates: First submitted 2013-03-11; First posted 2013-05-03 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Hypoventilation
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non invasive ventilation

SUMMARY:
The purpose of this study is to determine whether clinical examination, report from ventilator software, nocturnal Sp02 and daytime arterial blood gas are sufficient as screening tools to reveal clinical relevant problems with patients receiving long term treatment with non invasive ventilation.

DETAILED DESCRIPTION:
Patient with chronic hypoventilation with stable on long term treatment (LTMV) with non-invasive ventilation for at least 3 month taking part of our LTMV program will be included.

In addition to clinical examination,report from ventilator software, nocturnal Sp02 and daytime arterial blood gas all patients will be investigated with sleep polygraphy and transcutaneous Co2.

ELIGIBILITY:
* Admitted to our unit for optimal treatment of long term non invasive ventilation
* Readmitted for control after 6-8 weeks
* Then treated for at least 3 month with long term non invasive ventilation outside of hospital.
* Informed written consent

Exclusion Criteria:

* Under 18 years old
* Lack of cooperation
* Pregnant
* Acute exacerbation last 3 month leading to hospital admission.
* Change of treatment last 3 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hypoventilation treated with long term mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Frequency of transcutaneous co2 revealing sleep hypoventilation, when nocturnal pulseoximeter is normal | single night study

SECONDARY OUTCOMES:
Frequency of patient-ventilator asynchrony during non invasive ventilation ? | Single night study

OTHER OUTCOMES:
Technical drift of Transcutaneous Co2 measurement during 8 hours monitoring | One night study
Interscorer variability when scoring polygraphy during Non invasive ventilation | one night study
Comparing rate of event data from ventilator software with manually scored polygraphy during non invasive ventilation | Single night study
Accuracy of Transcutaneous monitoring of Co2 compared to arterial carbon dioxide partial pressure | single night study
Frequency of sleep related breathing events during non invasive ventilation | single night study

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd aarrestad, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Aarrestad S, Qvarfort M, Kleiven AL, Tollefsen E, Skjonsberg OH, Janssens JP. Diagnostic accuracy of simple tools in monitoring patients with chronic hypoventilation treated with non-invasive ventilation; a prospective cross-sectional study. Respir Med. 2018 Nov;144:30-35. doi: 10.1016/j.rmed.2018.09.015. Epub 2018 Sep 26. PMID 30366581
- [Derived] Aarrestad S, Qvarfort M, Kleiven AL, Tollefsen E, Skjonsberg OH, Janssens JP. Sleep related respiratory events during non-invasive ventilation of patients with chronic hypoventilation. Respir Med. 2017 Nov;132:210-216. doi: 10.1016/j.rmed.2017.10.025. Epub 2017 Nov 2. PMID 29229100
- [Derived] Aarrestad S, Tollefsen E, Kleiven AL, Qvarfort M, Janssens JP, Skjonsberg OH. Validity of transcutaneous PCO2 in monitoring chronic hypoventilation treated with non-invasive ventilation. Respir Med. 2016 Mar;112:112-8. doi: 10.1016/j.rmed.2016.01.017. Epub 2016 Jan 27. PMID 26874895